CLINICAL TRIAL: NCT02730481
Title: A Dose Regimen-Finding Study to Evaluate the Safety, Tolerability, Maximum Tolerated Dose, Pharmacokinetics, and Activity of Oraxol in Subjects With Advanced Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability, MTD, PK, and Activity of Oraxol in Subjects w Adv. Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-004
Record Dates: First submitted 2016-03-03; First posted 2016-04-06 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ORAXOL (Experimental): Oraxol (paclitaxel + HM30181AK-US) Oraxol paclitaxel - supplied as 30-mg capsules
  Oraxol HM30181 methanesulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — Oraxol will be supplied as paclitaxel capsules and HM30181AK-US tablets.
  Other Names: Paclitaxel and HM30181AK-US

SUMMARY:
This is a multicenter, open-label, safety study. Eligible subjects will be adults with advanced malignancies. The study includes a pretreatment and treatment phase. The pretreatment phase consists of screening and baseline periods. The treatment phase consists of 4-week treatment periods and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. ≥18 years of age
3. Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
4. Measurable disease as per RECIST v1.1 criteria
5. Adequate hematologic status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain: ANC ≥1500 cells/mm3, Platelet count ≥100 x 109/L, Hemoglobin ≥9 g/dL
6. Adequate liver function as demonstrated by:Total bilirubin of ≤1.5 mg/dL or ≤2.0 mg/dL for subjects with liver metastasis, Alanine aminotransferase ≤3 x upper limit of normal (ULN) or ≤5 x ULN if liver metastasis is present, Alkaline phosphatase ≤3 x ULN or ≤5 x ULN if bone or liver metastasis is present
7. Adequate renal function as demonstrated by serum creatinine ≤1.5 x ULN or creatinine clearance calculation ≥60 mL/min as calculated by the Cockcroft and Gault formula
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
9. Life expectancy of at least 3 months
10. Women must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of study drug.
11. Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.

Exclusion Criteria:

1. Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational products (IPs)
2. Received IPs within 30 days or 5 half lives of the first study dosing day
3. Are currently receiving other medications or radiation intended for the treatment of their malignancy
4. Women of childbearing potential who are pregnant or breastfeeding
5. Currently taking a concomitant medication
6. Require therapeutic use of anticoagulation medications
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements
8. Major surgery to the upper gastrointestinal (GI) tract, or have a history of GI disease or other medical condition that, in the opinion of the investigator may interfere with oral drug absorption
9. History of hypersensitivity to paclitaxel, not attributed to a hypersensitivity type reaction to Cremophor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Oraxol | 20 weeks
  The highest dose at which no more than 1 of 6 subjects experience a dose-limiting toxicity (DLT) during treatment

SECONDARY OUTCOMES:
Evaluate tumor response | At baseline and every 8 weeks through study completion, approximately 24 months
  RECIST v1.1 criteria defined as complete response, partial response, stable disease or progressive disease
Number of Participants with abnormal laboratory values and/or adverse events that are related to treatment | 4 weeks
  Number of Participants with abnormal laboratory values and/or adverse events that are related to treatment
The amount of Oraxol in the blood stream | 3 weeks
  The measurement of Oraxol levels in the blood stream over time
The recommended Phase 2 dose of paclitaxel as Oraxol | 24 months
  The totality of information from the number of participants that reach the MTD (outcome #1), the number of participants that experience abnormal laboratory values and/or adverse events that are related to treatment (outcome #3), and the amount of Oraxol in the blood stream in participants (outcome #4)

CONTACTS AND LOCATIONS:
Overall Officials: E D Kramer, MD, Study Director — Kinex Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cancer Therapy &Research Center @ UTHSCSA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No